CLINICAL TRIAL: NCT03091855
Title: Overall and MRI-based Impact of Percutaneous Left Atrial Appendage Closure on the Cognitive Decline and Dementia in Patients With Atrial Fibrillation (PLUG Dementia Trial and MRI PLUG Dementia Sub-Study)
Brief Title: PLUG Dementia Trial and MRI PLUG Dementia Sub-Study
Status: Terminated | Type: Observational
Why Stopped: Terminated due to low enrollment
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1050344
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation; Dementia; Cognitive Decline
MeSH Terms: conditions — Atrial Fibrillation; Dementia; Cognitive Dysfunction | interventions — Surveys and Questionnaires; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLUG Dementia Trial: Patients with atrial fibrillation that undergo a standard of care, clinically approved, left atrial appendage closure will be considered for study. All patients will be followed for 24 months, and will be assessed at the 3-, 6-, 12-, 18- and 24-months post-left atrial appendage closure as well as other visits deemed necessary for clinical care. All subjects will undergo protocol-specified laboratory tests and will complete 6 standard, validated questionnaires at each follow-up visit, except at the 3-month visit when only one questionnaire will be administered.
  Interventions: Other: Questionnaire
- MRI PLUG Dementia Sub-Study: 20 of the 60 subjects who are selected for participation in this sub-study will receive a cranial MRI at baseline and at the 2-year (24 months) follow-up visit.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Questionnaire — Alzheimer's Disease Assessment Scale (ADAS-cog11) and Disability Assessment for Dementia (DAD) Questionnaires
  Groups: PLUG Dementia Trial
Diagnostic Test: Magnetic Resonance Imaging — MRI at baseline and at 24 months post-enrollment for 20 sub-study participants
  Groups: MRI PLUG Dementia Sub-Study

SUMMARY:
PLUG Dementia Trial:

Patients will be screened at Intermountain Medical Center and at Intermountain affiliated anticoagulation clinics in the Salt Lake City region. Patients with atrial fibrillation that undergo a standard of care, clinically approved, left atrial appendage closure will be considered for study. All patients will be followed for 24 months, and will be assessed at the 3-, 6-, 12-, 18- and 24-months post-left atrial appendage closure as well as other visits deemed necessary for clinical care. All subjects will undergo protocol-specified laboratory tests and will complete 6 standard, validated questionnaires at each follow-up visit, except at the 3-month visit when only one questionnaire will be administered. A subset of patients (n=20), will receive a cranial MRI at baseline and 24-month visit.

MRI PLUG Dementia Sub-Study:

In addition to the above, 20 of the 60 subjects who are selected for participation in this sub-study will receive a cranial MRI at baseline and at the 2-year (24 months) follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >65 years of age
2. Atrial fibrillation documented by electrocardiogram, ambulatory event monitor, or telemetry within 6 months of enrollment
3. Moderate risk of thromboembolism based upon a CHADS2 score or CHADS2 Vasc score of ≥2.
4. Recipient of a left atrial appendage closure device within 3 months of enrollment (within 6 months, for patients considered for the MRI PLUG Dementia Sub-Study)
5. Have the ability to complete a mini-mental status evaluation
6. Have the ability to independently comprehend and complete a quality of life and dementia questionnaires.
7. Ability to provide informed consent for study participation
8. Willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

1. Have a history of any form of dementia
2. Have a life expectancy less than 24 months
3. Are unable to comply with the follow-up schedule
4. An upper age limit not to be used if participation inclusion criteria are met.
5. Participation in any other clinical trials involving an investigational or marketed drug within 30 days prior to entry in this study;
6. Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial
7. The Principal Investigator(s) determine(s) that the subject is not eligible for participation in this research study.

In addition to the above exclusion criteria, patients considered for the MRI PLUG Dementia Sub-Study will be excluded if the patient -

1. Does not receive a left atrial appendage closure device
2. Has contraindication towards the MRI scan (presence of a nonconditional cardiac implantable device, a history of metallic implants, shrapnel, neurosurgical clip placement)
3. Has conditional cardiac MRI cardiac implantable device, joint replacements, coronary stents, ASD/PFO closure devices, sternal wires or most prosthetic heart valves
4. Has severe renal dysfunction, defined as a creatinine clearance <15 mL/min (documented within the last 3 months)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with atrial fibrillation that undergo a standard of care, clinically approved, left atrial appendage closure will be considered for study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Dementia Incidence | 24 months
  Incident dementia determined by a formal diagnosis by a neurologist.
Change in cognitive decline | 24 months
  Moderate cognitive decline defined as a 30% decrease in Alzheimer's Disease Assessment Scale score or those with a score <50% or a 30% change on the Disability Assessment for Dementia.
Incidence of baseline micro- and macro-cerebral ischemic events (Sub-study Participants) | 24 months
  assess the incidence of baseline micro- and macro-cerebral ischemic events (both bleeds and clots) at the time of left atrial appendage closure and compare this with a serial study.

SECONDARY OUTCOMES:
Changes in cranial MRI | 24 months
  Incidence of bleeding and/or clots in the brain.

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Heart Institute, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No